CLINICAL TRIAL: NCT05615051
Title: Influence of Implant Surface Decontamination on the Reconstructive Outcomes of Peri-implantitis: A Randomized Clinical Trial
Brief Title: Influence of Implant Surface Decontamination on the Reconstructive Outcomes of Peri-implantitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31102022
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group electrolytic approach (EA) (Experimental): Mechanical detoxification using curettes + NiTi brushes + EA (GalvoSurge) during 2 minutes
  Interventions: Device: Surface decontamination procedure aiming at reconstructive therapy
- Group hydrogen peroxide (HP) (Active Comparator): Group hydrogen peroxide (HP): Mechanical detoxification using curettes + NiTi brushes + hydrogen peroxide 5% for 2 minutes soaked in a gauze
  Interventions: Device: Surface decontamination procedure aiming at reconstructive therapy

INTERVENTIONS:
Device: Surface decontamination procedure aiming at reconstructive therapy — Surface decontamination of infected implants followed by reconstructive therapy to manage peri-implantitis
  Other Names: Hydrogen peroxide

SUMMARY:
Two groups are aimed at being investigated in three centers (CICOM, Clinica Branemark and Clinica Joan Pi)

* Test group: Group electrolytic approach (EA): Mechanical detoxification using curettes + NiTi brushes + EA (GalvoSurge) during 2 minutes
* Control group: Group hydrogen peroxide (HP): Mechanical detoxification using curettes + NiTi brushes + hydrogen peroxide 5% for 2 minutes soaked in a gauze Patients´ group selection will be randomly allocated. For patients whom their personal clinical record # ends in a number from 0 to 4 will be included in the test group, while for patients whom their personal clinical record # ends from 5-9 will be included in the control group.

The infra-osseous component will be regenerated using xenograft (Creos, NB) + autogenous bone in a ratio 1:1 harvested from the adjacent area. A resorbable membrane (Creos, NB) will be placed to compartmentalize the infra-osseous component following a poncho-like approach.

ELIGIBILITY:
Inclusion:

* Screw-retained or cement-retained fixed or removable implant-supported prosthesis for a minimum of 36 months.
* All patients in age of 18 to 80
* non-smokers
* no presence of systemic disease or medication known to alter bone metabolism
* partial or complete edentulous patients that have no active periodontal disease.

Exclusion criteria:

* pregnancy or lactation
* history of or current smokers
* uncontrolled medical conditions,
* lacking keratinized mucosa (≤2mm) on the lingual or buccal implant sites,
* advanced(A) peri-implantitis (>50% of the implant length).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Resolution of the disease | 12 months
  No pocket depth >6mm, no bleeding on probing, no suppuration, no progressive bone loss

SECONDARY OUTCOMES:
Radiographic bone gain and clinical outcomes | 12 months
  Bone gain and changes in defect angle when compared to baseline radiographic features and evolution of clinical parameters compared to baseline data

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica CICOM, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monje A, Navarro-Mesa S, Soldini C, Zappala G, Pena P, Navarro JM Sr, Pons R. Surface Decontamination on the Reconstructive Therapy of Peri-Implantitis: A Multicenter Randomized Clinical Trial. Clin Implant Dent Relat Res. 2025 Aug;27(4):e70075. doi: 10.1111/cid.70075. PMID 40693504